CLINICAL TRIAL: NCT06899191
Title: Diabetes Electronic Prompt for Improved Care Coordination and Treatment (DEPICCT) in the ED
Brief Title: Diabetes Electronic Prompt for Improved Care Coordination and Treatment in the ED
Acronym: DEPICCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Paul Peng, MD PhD MSCR, Assistant Professor, Rutgers, The State University of New Jersey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Pro2024002629
Record Dates: First submitted 2025-03-21; First posted 2025-03-27 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Type 2 Diabetes; Type 2 Diabetes Mellitus (T2DM); Hyperglycemia; Insulin Dependent Diabetes
Keywords: Type 2 Diabetes; Electronic Prompt; Emergency Department Diabetes; Practice Advisory
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hyperglycemia; Diabetes Mellitus, Type 1 | interventions — Clinical Observation Units

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental): All ED providers exposed to electronic alerts
  Interventions: Diagnostic Test: Hemoglobin A1c; Behavioral: Observation Unit

INTERVENTIONS:
Diagnostic Test: Hemoglobin A1c — Prompt to order A1c
Behavioral: Observation Unit — Electronic prompt nudging ED provider to consider admitting patient to the Observation Unit for care coordination and more aggressive glycemic control

SUMMARY:
The goal of this clinical trial is to improve the processes of Type 2 Diabetes (T2D) care coordination and treatment in the emergency department (ED) by utilizing clinical decision support mechanisms in the electronic health record (EHR). The main question is whether electronic prompts triggered by hyperglycemia and elevated A1c results in providers providing earlier treatments and faster time to subsequent primary care appointment and greater reduction in hemoglobin A1c (HA1c).

ED clinicians will receive alerts called Our Practice Advisories (OPA's) through the EPIC EHR. The 1st OPA triggers when a random point-of-care (POC) glucose is ≥250 mg/dL, prompting a suggested additional HA1c order. A 2nd OPA triggers if the resulting HA1c is ≥10%, prompting consideration of further care coordination in the Observation Unit. Investigators will compare the outcomes post-intervention compared to pre-intervention.

DETAILED DESCRIPTION:
Type 2 Diabetes (T2D) is a growing public health crisis with rates of diabetes steadily increasing over the last 10 years. The ED is commonly the first point of contact for individuals who present with symptoms of hyperglycemia, often with very severe (HbA1C > 10%) underlying diabetes. However, there is currently no national guideline or clinical policy for the ED management of patients who are not in diabetic ketoacidosis (DKA) or in a hyperglycemia hyperosmolar state (HHS). The investigators hypothesize that there are two subgroups who may benefit from greater care coordination initiated from the ED: patients who are newly-diagnosed with severe T2D and patients whom T2D is poorly-controlled despite medication adherence. This study designs electronic prompt practice advisories that nudge ED providers towards more aggressive treatment pathways. It is currently unknown whether alert tools can improve the delivery and coordination of care of patients with severe T2D presenting to the ED.

ELIGIBILITY:
Inclusion Criteria:

Moderate hyperglycemia, (glucose ≥250 mg/dL)

* Patients who arrive in the emergency department
* Not pregnant or peri-partum
* Not SARS-COV-2 PCR positive in past 7 days

Exclusion Criteria:

* Diabetic ketoacidosis (pH < 7.20, HCO3 < 15, AG > 25)
* Diabetic foot ulcer or skin complications
* Hyperglycemic hyperosmolar state with neurologic impairment
* Patients who leave against medical advice (AMA), elope from the ED, or are transferred to another facility

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-03-30 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Care Coordination: Follow-Up Care | From date of ED encounter until 4 weeks after
  % Patients achieving: A T2D-related appointment within 4 weeks
Physiologic Response | From date of ED encounter to 4 months after
  % Patients achieving: HbA1c 1% reduction in 3 months

SECONDARY OUTCOMES:
Care Coordination: Disposition | Within 1 day of ED encounter date
  number of patients discharged, number of patients admitted to observation unit, number of patients admitted to hospital
Care Coordination: Length of stay | 1 day
  Length of stay (minutes) of subject ED encounter
Care Coordination: Insurance | Within 3 weeks of ED encounter
  Inclusion: patients with NO insurance Measure % Patients achieving new insurance
Care Coordination: Medication Prescription | 3 days
  Inclusion: patients discharged from the ED or observation Unit
  % subjects prescribed a diabetes medication
Care Coordination: Medication Change | 3 days
  Inclusion: patients discharged from the ED or observation Unit
  % subjects with a change in diabetes medication regimen
Care Coordination: Appointment | 3 months
  Time (days) to next appointment related to T2D, calculated as [Appt date] - [ED encounter date]
Physiologic: A1c Orders | 1 day
  Proportion of patients with hemoglobin A1c ordered in the ED
Physiologic: Serum Glucose | 1 day
  Serum glucose concentration change from beginning to end of ED encounter
Physiologic: Hemoglobin A1c percentage | 6 months
  Serum hemoglobin A1c (%)
Physiologic: Diagnosis | 1 day
  Proportion of subjects with newly diagnosed Type 2 Diabetes, proportion of subjects with poorly controlled, established Type 2 Diabetes
Physiologic: ED medications | 1 day
  % subjects receiving (1) intravenous fluids, (2) insulin, (3) other diabetes medications while in the ED

CONTACTS AND LOCATIONS:
Locations (1):
- Rutgers, Robert Wood Johnson Hospital, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
Subject data stored on RedCap can be extracted with deidentified information for data sharing.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Until 1 year after study
Access Criteria: Only the Principal Investigator, PP, will have access
URL: https://research.rutgers.edu/faculty-staff/compliance/human-research-protection/clinical-trials

REFERENCES:
- [Background] Yan JW, Vujcic B, Le BN, Van Aarsen K, Chen T, Halane F, Clemens KK. Predictors of 30-day recurrent emergency department visits for hyperglycemia in patients with types 1 and 2 diabetes: a population-based cohort study. CJEM. 2024 Jun;26(6):424-430. doi: 10.1007/s43678-024-00686-4. Epub 2024 Apr 18. PMID 38635005
- [Background] Magee MF, Nassar C. Hemoglobin A1c testing in an emergency department. J Diabetes Sci Technol. 2011 Nov 1;5(6):1437-43. doi: 10.1177/193229681100500615. PMID 22226261
- [Background] Magee MF, Nassar CM, Copeland J, Fokar A, Sharretts JM, Dubin JS, Smith MS. Synergy to reduce emergency department visits for uncontrolled hyperglycemia. Diabetes Educ. 2013 May-Jun;39(3):354-64. doi: 10.1177/0145721713484593. Epub 2013 Apr 22. PMID 23610182
- [Background] King WM 4th, McDermott MT, Trujillo JM. Initial management of severe hyperglycemia in patients with type 2 diabetes: an observational study. Diabetes Ther. 2013 Dec;4(2):375-84. doi: 10.1007/s13300-013-0036-9. Epub 2013 Aug 16. PMID 23949906
- [Background] Ginde AA, Delaney KE, Pallin DJ, Camargo CA Jr. Multicenter survey of emergency physician management and referral for hyperglycemia. J Emerg Med. 2010 Feb;38(2):264-70. doi: 10.1016/j.jemermed.2007.11.088. Epub 2008 Jul 26. PMID 18657930
- [Background] Gale J, Varndell W, James S, Perry L. Unscheduled emergency department presentations with diabetes: Identifying high risk characteristics. Australas Emerg Care. 2023 Sep;26(3):205-210. doi: 10.1016/j.auec.2022.12.001. Epub 2022 Dec 15. PMID 36528482
- [Background] Driver BE, Olives TD, Prekker ME, Miner JR, Klein LR. The Association of Emergency Department Treatments for Hyperglycemia with Glucose Reduction and Emergency Department Length of Stay. J Emerg Med. 2017 Dec;53(6):791-797. doi: 10.1016/j.jemermed.2017.08.068. Epub 2017 Oct 6. PMID 28993036
- [Background] Driver BE, Olives TD, Bischof JE, Salmen MR, Miner JR. Discharge Glucose Is Not Associated With Short-Term Adverse Outcomes in Emergency Department Patients With Moderate to Severe Hyperglycemia. Ann Emerg Med. 2016 Dec;68(6):697-705.e3. doi: 10.1016/j.annemergmed.2016.04.057. Epub 2016 Jun 25. PMID 27353284
- [Background] Driver BE, Klein LR, Cole JB, Prekker ME, Fagerstrom ET, Miner JR. Comparison of two glycemic discharge goals in ED patients with hyperglycemia, a randomized trial. Am J Emerg Med. 2019 Jul;37(7):1295-1300. doi: 10.1016/j.ajem.2018.09.053. Epub 2018 Oct 5. PMID 30316635
- [Background] Davies MJ, Aroda VR, Collins BS, Gabbay RA, Green J, Maruthur NM, Rosas SE, Del Prato S, Mathieu C, Mingrone G, Rossing P, Tankova T, Tsapas A, Buse JB. Management of hyperglycaemia in type 2 diabetes, 2022. A consensus report by the American Diabetes Association (ADA) and the European Association for the Study of Diabetes (EASD). Diabetologia. 2022 Dec;65(12):1925-1966. doi: 10.1007/s00125-022-05787-2. Epub 2022 Sep 24. PMID 36151309
- [Background] Crawford AL, Laiteerapong N. Type 2 Diabetes. Ann Intern Med. 2024 Jun;177(6):ITC81-ITC96. doi: 10.7326/AITC202406180. Epub 2024 Jun 11. PMID 38857502
- [Background] Charfen MA, Ipp E, Kaji AH, Saleh T, Qazi MF, Lewis RJ. Detection of undiagnosed diabetes and prediabetic states in high-risk emergency department patients. Acad Emerg Med. 2009 May;16(5):394-402. doi: 10.1111/j.1553-2712.2009.00374.x. Epub 2009 Mar 16. PMID 19302369
- [Background] Bowen ME, Xuan L, Lingvay I, Halm EA. Random blood glucose: a robust risk factor for type 2 diabetes. J Clin Endocrinol Metab. 2015 Apr;100(4):1503-10. doi: 10.1210/jc.2014-4116. Epub 2015 Feb 4. PMID 25650899
- [Background] American Diabetes Association Professional Practice Committee. 2. Diagnosis and Classification of Diabetes: Standards of Care in Diabetes-2024. Diabetes Care. 2024 Jan 1;47(Suppl 1):S20-S42. doi: 10.2337/dc24-S002. PMID 38078589